CLINICAL TRIAL: NCT02791191
Title: Effect of LY3202626 on Alzheimer's Disease Progression as Measured by Cerebral ¹⁸F-AV-1451 Tau-PET in Mild Alzheimer's Disease Dementia
Brief Title: A Study of LY3202626 on Disease Progression in Participants With Mild Alzheimer's Disease Dementia
Acronym: NAVIGATE-AD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low likelihood of identifying a statistically significant treatment effect.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16223; I7X-MC-LLCF (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer's Disease
Keywords: BACE inhibitor
MeSH Terms: conditions — Alzheimer Disease | interventions — LY3202626

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 LY3202626 (Experimental): 3 mg LY3202626 given orally once daily for 52 weeks.
  Interventions: Drug: LY3202626
- Dose 2 LY3202626 (Experimental): 12 mg LY3202626 given orally once daily for 52 weeks.
  Interventions: Drug: LY3202626
- Placebo (Experimental): Placebo given orally once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3202626 — Administered orally
  Arms: Dose 1 LY3202626; Dose 2 LY3202626
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and the effect on brain tau of the study drug LY3202626 in participants with mild Alzheimer's disease (AD) dementia.

ELIGIBILITY:
Inclusion Criteria:

* Present with mild AD dementia based on the National Institute on Aging (NIA) and the Alzheimer's Association (AA) disease diagnostic criteria as determined by a qualified clinician approved by the Sponsor or designee.
* Mini-Mental State Examination score of 20 to 26 inclusive at screening visit.
* Has a florbetapir PET scan consistent with the presence of amyloid pathology at screening.

Exclusion Criteria:

* Significant neurological disease affecting the central nervous system (CNS), other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson's disease, multiple concussions, or epilepsy or recurrent seizures (except febrile childhood seizures).
* Ocular pathology that significantly limits ability to reliably evaluate vision or the retina.
* Use of strong inducers of cytochrome P450 3A (CYP3A).
* Sensitivity to florbetapir or ¹⁸F-AV-1451.
* Contraindication to MRI or PET or poor venous access for blood draws.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (75):
- United States (49):
  - Irvine Clinical Research Center, Irvine, California
  - Sutter Medical Group, Sacramento, California
  - Pacific Research Network Inc, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Ray Dolby Brain Health Center/Sutter Health/CPMC, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - North Bay Neuroscience Institute, Sebastopol, California
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Christiana Care Health Service, Wilmington, Delaware
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Compass Research, Melbourne, Florida
  - Florida International Research Center, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - The Neurology Research Group, LLC, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Meridien Research, Spring Hill, Florida
  - Axiom Research, Tampa, Florida
  - United Osteoporosis Center, Gainesville, Georgia
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Center for Memory, Newton, Massachusetts
  - Missouri Memory Center, Bolivar, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - Millenium Psychiatric Associates LLC, Creve Coeur, Missouri
  - St Lukes Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Pyramid Clinical Research, Monroe, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Dent Neurological Institute, Amherst, New York
  - Valley Medical Primary Care, Centerville, Ohio
  - University of Cincinnati Health Neurology, Dayton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Insight Clinical Trials, Shaker Heights, Ohio
  - Abington Neurological Associates, Abington, Pennsylvania
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Trial Center, LLC, Psychiatry, Jenkintown, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Baylor AT&T Memory Center, Dallas, Texas
  - Nantz National Alzheimer Center, Houston, Texas
  - University of Texas Health Services Center - Houston, Houston, Texas
- Australia (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chermside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darlinghurst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Iris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Perth
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gatineau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verdun
- Japan (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akashi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hachiōji
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ikeda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kasukabe-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nerima-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Setagaya-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takamatsu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wako
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yokosuka-shi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: Click here for more information about this study: A Study of LY3202626 on Disease Progression in Participants With Mild Alzheimer's Disease Dementia (NAVIGATE-AD) — http://www.lillytrialguide.com/en-US/studies/mild-alzheimer's%20disease/LLCF#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 mg LY3202626: 3 mg LY3202626 administered orally once daily for 52 weeks.
- 12 mg LY3202626: 12 mg LY3202626 administered orally once daily for 52 weeks.
- Placebo: Placebo administered orally once daily for 52 weeks.
Period: Overall Study
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Started | 55 | 128 | 133
Received One Dose of Study Drug | 55 | 127 | 133
Completed | 17 | 17 | 13
Not Completed | 38 | 111 | 120
Not completed — Adverse Event | 2 | 4 | 5
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Study Drug Non-Compliance | 0 | 2 | 0
Not completed — Site Closed by Sponsor | 1 | 1 | 3
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 29 | 101 | 109
Not completed — Withdrawal by Subject | 3 | 1 | 3
Not completed — Subject Withdrew Caregiver Circumstances | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo | Total
Number analyzed (Participants) | 55 | 128 | 133 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.91 (6.72) | 72.73 (7.15) | 72.54 (7.80) | 72.86 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 86 | 77 | 192
  Male | 26 | 42 | 56 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 7 | 13
  Not Hispanic or Latino | 50 | 108 | 112 | 270
  Unknown or Not Reported | 4 | 15 | 14 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 18 | 13 | 39
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 1 | 5 | 4 | 10
  White | 45 | 104 | 113 | 262
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 1 | 2
  United States | 43 | 86 | 105 | 234
  Japan | 7 | 18 | 12 | 37
  Australia | 5 | 23 | 15 | 43
Flortaucipir Standard Uptake Value Ratio (SUVr) [Mean (Standard Deviation); unit: standard uptake value ratio (SUVr)] — Population: Participants who completed the baseline ¹⁸F-AV-1451 Positron Emission Tomography (PET) and had evaluable Standard Uptake Value Ratio (SUVr).
  standard uptake value ratio (SUVr)
    number analyzed (Participants) | 52 | 121 | 119 | 292
    (all) | 1.32 (0.24) | 1.36 (0.28) | 1.42 (0.35) | 1.38 (0.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ¹⁸F-AV-1451 Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVr) at 52 Weeks
Description: The 18F-AV-1451 PET tracer assesses change from baseline in the pharmacodynamic effect of 3 mg and 12 mg doses of LY3202626 in participants with mild Alzheimer's disease (AD), compared with placebo at Week 52.The SUVr of ¹⁸F-AV-1451 was modeled using analysis of covariance (ANCOVA) to include the fixed, categorical effects of treatment dose, and the continuous, fixed covariate of baseline Tau PET SUVr and age at baseline.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug, and have baseline and at least one post-baseline scan.
Measure: Mean (Standard Deviation); unit: Standard Uptake Value Ratio (SUVr)
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 15 | 15 | 11
Standard Uptake Value Ratio (SUVr) | 0.02 (0.04) | 0.03 (0.04) | 0.01 (0.08)
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.418, ANCOVA
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.231, ANCOVA

2. Secondary Outcome: Percentage of Participants With Emergent Magnetic Resonance Imaging (MRI) Findings
Description: Percentage of participants with treatment-emergent MRI findings at Week 52 are summarized here. The mixed-effect model for repeated measures (MMRM) analysis was adjusted for fixed effects of treatment, visit (categorical covariate), treatment-by-visit interaction, baseline age, baseline score (continuous covariate) and baseline-by-visit interaction.
Time Frame: Week 52
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 41 | 75 | 62
percentage of participants
  White Matter Disease | 2.4 | 1.3 | 1.6
  Cortical Infarct | 2.4 | 0.0 | 0.0
  Cortical Superficial Siderous | 0.0 | 1.3 | 0.0
  Lacunar Infarct | 0.0 | 0.0 | 1.6
  Other Infarct | 0.0 | 0.0 | 1.6
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; White Matter Disease; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; White Matter Disease; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: 3 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.404, Fisher Exact
Statistical Analysis 4: Comparison: 12 mg LY3202626 vs Placebo; Cortical Superficial Siderous; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 5: Comparison: 3 mg LY3202626 vs Placebo; Test type: Superiority — Lacunar Infarct; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: 12 mg LY3202626 vs Placebo; Lacunar Infarct; Test type: Superiority; p = 0.457, Fisher Exact
Statistical Analysis 7: Comparison: 3 mg LY3202626 vs Placebo; Other Infarct; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 8: Comparison: 12 mg LY3202626 vs Placebo; Other Infarct; Test type: Superiority; p = 0.457, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Amyloid-Related Imaging Abnormalities (ARIA)
Description: Percentage of participants with presence of amyloid-related imaging abnormalities-edema (ARIA-E, also known as vasogenic edema) and percentage of an increase in amyloid-related imaging abnormalities-hemorrhage (ARIA-H, also known as also known as microhemorrhage) at Week 52 are summarized here. The mixed-effect model for repeated measures (MMRM) analysis was adjusted for fixed effects of treatment, visit (categorical covariate), treatment-by-visit interaction, baseline age, baseline score (continuous covariate) and baseline-by-visit interaction.
Time Frame: Week 52
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 41 | 75 | 62
percentage of participants
  Presence of Vasogenic Edema | 0.0 | 0.0 | 1.6
  Increase in Microhemorrhages | 4.7 | 6.3 | 7.5
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Vasogenic Edema; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Vasogenic Edema; Test type: Superiority; p = 0.457, Fisher Exact
Statistical Analysis 3: Comparison: 3 mg LY3202626 vs Placebo; Increase in Microhemorrhage; Test type: Superiority; p = 0.703, Fisher Exact
Statistical Analysis 4: Comparison: 12 mg LY3202626 vs Placebo; Increase in Microhemorrhage; Test type: Superiority; p = 1.000, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Suicidal Ideation and Behaviors Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Scores
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation is defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which includes a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation and behavior are defined as treatment-emergent (TE) if not present during the period up through randomization. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through Week 52
Population: All participants who received at least one dose of study drug and had at least one post-baseline C-SSRS measure.
Measure: Number; unit: percentage of participants
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 55 | 127 | 133
percentage of participants
  TE Suicidal Ideation | 7.27 | 7.09 | 3.76
  TE Suicidal Behavior: number analyzed (Participants) | 55 | 126 | 133
  TE Suicidal Behavior | 1.82 | 0.79 | 0.00
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Treatment Emergent Suicidal Ideation; Test type: Superiority; p = 0.452, Fisher Exact
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.279, Fisher Exact — TE Suicidal Ideation
Statistical Analysis 3: Comparison: 3 mg LY3202626 vs Placebo; Emergence of Suicidal Behavior; Test type: Superiority; p = 0.293, Fisher Exact
Statistical Analysis 4: Comparison: 12 mg LY3202626 vs Placebo; Emergence of Suicidal Behavior; Test type: Superiority; p = 0.486, Fisher Exact

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve at Steady State (AUC [T,SS]) of LY3202626
Description: PK: AUC [T,SS] of LY3202626
Time Frame: Week 2, 4, and 12: Predose and Postdose prior to departing; Week 8 and 16: Postdose after arriving and prior to departing; Week 24: Postdose after cognitive testing
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626
Number analyzed (Participants) | 55 | 127
nanogram*hour per milliliter (ng*h/mL) | 158 (55.1) | 641 (58.0)

6. Secondary Outcome: Change From Baseline in Plasma Amyloid Beta Aβ₁-₄₀, ₁-₄₂, and 1-x Concentration
Description: A mixed model repeated measures (MMRM) analysis will be used to evaluate the change from baseline to Week 52 in plasma Aβ₁-₄₀, Aβ₁-₄₂, and Aβ 1-x. The model for the fixed effects will include terms for the following independent effects: log transformed baseline plasma Aβ, treatment, visit, treatment-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug, and have baseline and at least one post-baseline measure.
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 55 | 127 | 133
nanograms per liter (ng/L)
  Amyloid Beta: number analyzed (Participants) | 13 | 17 | 14
  Amyloid Beta | -258.7 (64) | -286.1 (85.9) | -12.0 (80.5)
  Amyloid Beta 1-40: number analyzed (Participants) | 14 | 17 | 15
  Amyloid Beta 1-40 | -157.3 (65.6) | -149.3 (38.0) | -17.0 (38.2)
  Amyloid Beta 1-42: number analyzed (Participants) | 14 | 17 | 15
  Amyloid Beta 1-42 | -46.3 (38.7) | -50.0 (34.1) | 0.0 (5.8)
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Amyloid Beta; Test type: Superiority; p < .001, ANCOVA
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Test type: Superiority — Amyloid Beta; p < .001, ANCOVA
Statistical Analysis 3: Comparison: 3 mg LY3202626 vs Placebo; Amyloid Beta 1-40; Test type: Superiority; p < .001, ANCOVA
Statistical Analysis 4: Comparison: 12 mg LY3202626 vs Placebo; Amyloid Beta 1-40; Test type: Superiority; p < .001, ANCOVA
Statistical Analysis 5: Comparison: 3 mg LY3202626 vs Placebo; Amyloid Beta 1-42; Test type: Superiority; p < .001, ANCOVA
Statistical Analysis 6: Comparison: 12 mg LY3202626 vs Placebo; Amyloid Beta 1-42; Test type: Superiority; p < .001, ANCOVA

7. Secondary Outcome: Change From Baseline on the 13-item Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog₁₃)
Description: The ADAS is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS that was used as the primary efficacy measure consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS--Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. A mixed model repeated measures (MMRM) was used in analysis. The model included fixed, categorical effects of treatment, visit and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline, baseline-by-visit, and age at baseline.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug, and have baseline and at least one post-baseline ADAS-Cog₁₃ measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 17 | 19 | 15
units on a scale | 3.05 (1.40) | 1.88 (1.33) | 2.97 (1.51)
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.970, Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.586, Mixed Model Repeated Meausres

8. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Inventory (ADCS-iADL)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities (instrumental activity items 7-23) of daily living by participants. The range for the ADCS-iADL is 0-56 with higher scores reflecting better performance. ADCS-iADL was analyzed using mixed-model repeated measures (MMRM), Least Square (LS) Mean was controlled for treatment, visit, treatment-by-visit interaction, baseline age, baseline score and baseline-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug, and have baseline and at least one post-baseline ADCS-iADL measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 17 | 19 | 15
units on a scale | -3.97 (1.34) | -4.63 (1.24) | -7.32 (1.38)
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.088, ANCOVA
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.150, ANCOVA

9. Secondary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS)
Description: The iADRS comprises scores form the ADAS-Cog and the ADCS-iADL. The iADRS is calculated as a linear combination of the total scores of the ADAS-Cog13 9score range 0 to 85 with higher scores reflecting worse performance and the ADCS-iADL (score range 0-56 with higher scores reflecting better performance). The iADRS score ranges from 0 to 141 with lower scores indicating worse performance. iADRS was analyzed using mixed-model repeated measures (MMRM); Least Square (LS) Mean was controlled for treatment, visit, treatment-by-visit interaction, baseline age, baseline score and baseline-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All participants who received at least one dose of study drug, and have baseline and at least one post-baseline iADRS measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
Number analyzed (Participants) | 16 | 19 | 15
units on a scale | -6.01 (2.07) | -6.45 (1.90) | -10.32 (2.15)
Statistical Analysis 1: Comparison: 3 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.153, ANCOVA
Statistical Analysis 2: Comparison: 12 mg LY3202626 vs Placebo; Test type: Superiority; p = 0.176, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to 56 Weeks
Description: All randomized participants.
Arm/Group | 3 mg LY3202626 | 12 mg LY3202626 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/127 | 0/133
Serious Adverse Events (participants affected / at risk) | 10/55 | 8/127 | 10/133
Other Adverse Events (participants affected / at risk) | 46/55 | 97/127 | 91/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg LY3202626 (N=55) | 12 mg LY3202626 (N=127) | Placebo (N=133)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg LY3202626 (N=55) | 12 mg LY3202626 (N=127) | Placebo (N=133)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 1 (1) | 1 (2)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dyschromatopsia (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Erythropsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lenticular opacities (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Normal tension glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Optic disc disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic disc haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal drusen (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (7) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Crying (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 5 (5) | 7 (7)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 6 (7) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 4 (5) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0)
Unevaluable event (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Mite allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Mycotic allergy (Immune system disorders) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Nail bed infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (7) | 14 (16) | 7 (7)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (6) | 7 (8)
Urinary tract infection (Infections and infestations) | 3 (5) | 7 (8) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 11 (12) | 4 (4)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 8 (12) | 8 (9)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Biopsy skin (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cystoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 3 (3) | 1 (1)
Fibrin d dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Mammogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 8 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint space narrowing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 4 (4)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Corticobasal degeneration (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 4 (4) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Superficial siderosis of central nervous system (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 3 (4) | 2 (2)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (4) | 3 (3) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (4)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 6 (6) | 2 (2)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0)
Hypnopompic hallucination (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 4 (5) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Idiopathic guttate hypomelanosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Leukoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3)
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Orthosis user (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Walking aid user (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Blepharectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bursa removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (3)
Catheter placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Chest tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cochlea implant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Lens capsulotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Micrographic skin surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nasal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Open reduction of fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Papilloma excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Vertebroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 5 (5) | 1 (1)
Supine hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated due to low likelihood of identifying a statistically significant treatment effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT02791191/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT02791191/SAP_001.pdf